CLINICAL TRIAL: NCT02856126
Title: The Efficacy and Safety of Hepatic Arterial Infusion Chemotherapy Plus Sorafenib Compared With Transarterial Chemoembolization Plus Sorafenib in Patients With BCLC C Stage Hepatocellular Carcinoma
Brief Title: HAIC Plus Sorafenib Versus TACE Plus Sorafenibfor Advanced HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S022
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic arterial infusion chemotherapy; Transarterial Chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HAIC plus sorafenib (Experimental): Procedure/Surgery: Hepatic arterial infusion chemotherapy Drug: HAIC Regimen Drug: Oral Sorafenib
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: HAIC Regimen; Drug: Oral Sorafenib
- TACE plus sorafenib (Active Comparator): Procedure/Surgery: Transarterial chemoembolization Drug: TACE regimen Drug: Oral Sorafenib
  Interventions: Procedure: Transarterial chemoembolization; Drug: TACE regimen; Drug: Oral Sorafenib

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy
  Arms: HAIC plus sorafenib
Procedure: Transarterial chemoembolization
  Arms: TACE plus sorafenib
Drug: TACE regimen — infusion with lipiodol mixed with chemotherapy drugs (EADM , lobaplatin, and MMC ), and embolization with polyvinyl alcohol particles (PVA)
  Arms: TACE plus sorafenib
Drug: HAIC Regimen — Hepatic intra-arterial infusion via the tumor feeding arteries of Oxaliplatin , fluorouracil, and leucovorin
  Arms: HAIC plus sorafenib
Drug: Oral Sorafenib — Oral Sorafenib, 400mg, Bid

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy (HAIC) compared with transarterial chemoembolization (TACE) in patients with BCLC stage hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) is the most widely used palliative treatment for hepatocellular carcinoma (HCC) patients. Our previous prospective study also revealed that TACE confers a survival benefit to patients with HCC and portal venous tumor thrombus (PVTT). Recently, the results of our preliminary pilot study suggested that, compared with TACE, hepatic arterial infusion chemotherapy (HAIC) may improve the survivals for patitens with BCLC stage C HCC. Thus, the investigators carried out this prospective randomized control study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of BCLC C stage HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* with no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

  * Platelet count ≥ 75,000/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 30mmol/L
  * Serum albumin ≥ 30 g/L
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or PT/APTT within normal limits
  * Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Main portal vein occlusion
* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | 18 months
  Overall survival

SECONDARY OUTCOMES:
Progress free survival | 18 months
  Progress free survival
Adverse Events | 30 Days
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v3.0
Number of of Patients developed Adverse Events | 30 Days
  Number of of patients who developed adverse event. Postoperative adverse events were graded based on CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — The Department of Hepatobiliary Oncology of Sun Yat-sen University Cancer Center
Locations (7):
- China (7):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospital, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong
  - The First Affiliated Hospital of University Of South China, Hengyang, Hunan
  - The First Affiliated Hospital Of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided